CLINICAL TRIAL: NCT03061071
Title: A Prospective, Randomized, Crossover Study of the NightBalance Sleep Position Trainer (SPT) Compared to Automatic Adjusting Positive Airway Pressure (APAP) for the Treatment of Positional Obstructive Sleep Apnea (POSA)
Brief Title: The POSAtive Study: Study for the Treatment of Positional Obstructive Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NightBalance (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: US-2017-001
Record Dates: First submitted 2017-02-13; First posted 2017-02-23 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Sleep Apnea Syndromes
Keywords: Positional Sleep Apnea; Positional Obstructive Sleep Apnea; POSA; OSA; Obstructive Sleep Apnea; Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: 6 week crossover study, randomized to order of treatment
Who Masked: Outcomes Assessor
Masking Description: The technician scoring the polysomnograms will be unaware of previous PSG results from the patient to the best of their ability (ie: will not look back in their records for the purpose of reviewing their previous PSGs prior to scoring).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Randomized to SPT First: APAP Second (Experimental): Randomized to order of treatment (SPT first or APAP first) for a total of 6 weeks home use with each treatment.
  Interventions: Device: NightBalance Sleep Position Trainer (SPT); Device: Automated Adjusting Positive Airway Pressure (APAP)
- Randomized to APAP First: SPT Second (Experimental): Randomized to order of treatment (APAP first or SPT first) for a total of 6 weeks home use with each treatment.
  Interventions: Device: NightBalance Sleep Position Trainer (SPT); Device: Automated Adjusting Positive Airway Pressure (APAP)

INTERVENTIONS:
Device: NightBalance Sleep Position Trainer (SPT) — Subject to sleep with the SPT for a 6 week home use period followed by in-lab PSG.
Device: Automated Adjusting Positive Airway Pressure (APAP) — Subject to sleep with the APAP for a 6 week home use period followed by in-lab PSG.

SUMMARY:
This study is a prospective, multi-center, randomized crossover of the NightBalance SPT compared to APAP for the treatment of Positional Obstructive Sleep Apnea (POSA).

DETAILED DESCRIPTION:
This study is a prospective, multi-center, randomized crossover of the NightBalance SPT compared to APAP for the treatment of POSA.

The Primary Objective of the study is to demonstrate non-inferiority of treatment with the SPT as compared to APAP.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is between the ages of 20 and 80.
2. Diagnosis of POSA meeting all the following criteria per in-lab control PSG (performed within 3 months of screening):

   * Total AHI >15, or AHI >10 and <15 with ESS >10
   * Supine AHI at least twice the non-supine AHI
   * Non-supine AHI <10 (<5 in mild patients)
   * Supine time >40% and <60%
3. Subject understands the study protocol and is willing and able to comply with study requirements and sign informed consent.

Exclusion Criteria:

1. Prior surgery to treat OSA (such as UPPP), or prior or current therapy or treatment for OSA, with the exception of PAP being used for split night PSG only.
2. A female of child-bearing potential that is pregnant or intends to become pregnant.
3. Any unstable or severe medical condition of any organ system including congestive heart failure, COPD, renal failure, neuromuscular disease, or at the discretion of the site Principal Investigator (PI).
4. Taking medication that may affect sleep, sleepiness, or alertness including hypnotics, sedatives, alerting agents, stimulants, opiates, sedating antidepressants, and anticonvulsants.
5. Oxygen use.
6. The presence of any other sleep disorder (central sleep apnea (CSA >5), periodic limb movement disorder (PLMAI >15), clinical diagnosis of insomnia or narcolepsy).
7. Excessive alcohol consumption (>21 drinks/week).
8. The use of any illegal drug(s).
9. Night or rotating shift work.
10. Severe claustrophobia.
11. Shoulder, neck, or back complaints that restrict sleeping position.
12. Subject requires use of more than 2 pillows under the head while sleeping or sleeps in a bed/chair with raised upper body position.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-07-12 (Actual)

PRIMARY OUTCOMES:
Adherence (minutes of device use per night) | 6 week
  Non-inferiority of SPT vs. APAP (calculated by number of minutes of objective device use per night)
Apnea-Hypopnea Index (AHI, events/hr) | 6 week
  Non-inferiority of SPT vs. APAP (measured by events/hr during in lab polysomnography)

SECONDARY OUTCOMES:
Epworth Sleepiness Scale (ESS) | 6 week
  SPT vs. APAP
Functional Outcomes of Sleep Questionnaire (FOSQ) | 6 week
  SPT vs. APAP
SF-36 | 6 week
  SPT vs. APAP
Patient Satisfaction (Comfort, Satisfaction) assessed by Visual Analog Scale (VAS) | 6 week
  SPT vs. APAP
Oxygen Desaturation Index (3%) | 6 week
  SPT vs. APAP
Total Sleep Time (minutes) | 6 week
  SPT vs. APAP (measured by in lab polysomnography)
Sleep Onset Latency (minutes) | 6 week
  SPT vs. APAP (measured by in lab polysomnography)
Sleep Efficiency (%) | 6 week
  SPT vs. APAP (measured by in lab polysomnography)
Arousal Index | 6 week
  SPT vs. APAP (measured by in lab polysomnography)
Sleep Stages (%) | 6 week
  SPT vs. APAP (measured by in lab polysomnography)
Sleep Position (%) | 6 week
  SPT vs. APAP (measured by in lab polysomnography)
Mean Disease Alleviation (MDA) (%) | 6 weeks
  SPT vs. APAP (MDA (%) is calculated by the product of the objective adherence (from SPT and APAP download), adjusted for total sleep time (X-axis), combined with therapeutic efficacy (AHI from the respective treatment night, Y-axis), divided by 100.)
Adverse Events | 6 weeks
  SPT vs. APAP, frequency, seriousness, severity and device relationship will be summarized.

CONTACTS AND LOCATIONS:
Overall Officials: Richard B Berry, MD, Principal Investigator — UF Health Sleep Center
Locations (11):
- United States (11):
  - Sleep Disorders Center of Alabama, Birmingham, Alabama
  - Sleep Med Inc., AZ, Glendale, Arizona
  - Sleep Disorders at Magnolia Park, Gainesville, Florida
  - Kentucky Research Group, Louisville, Kentucky
  - Center for Sleep and Wake Disorders, Chevy Chase, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - St. Luke's Sleep Medicine and Research Center, Chesterfield, Missouri
  - Clayton Sleep Institute, Maplewood, Missouri
  - Med One Sleep, Fayetteville, North Carolina
  - Pearl Clinical Research, Paoli, Pennsylvania
  - SleepMed of South Carolina, Columbia, South Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berry RB, Uhles ML, Abaluck BK, Winslow DH, Schweitzer PK, Gaskins RA Jr, Doekel RC Jr, Emsellem HA. NightBalance Sleep Position Treatment Device Versus Auto-Adjusting Positive Airway Pressure for Treatment of Positional Obstructive Sleep Apnea. J Clin Sleep Med. 2019 Jul 15;15(7):947-956. doi: 10.5664/jcsm.7868. PMID 31383231